CLINICAL TRIAL: NCT06768060
Title: Preparing Mothers for External Cephalic Version: a Mindfulness-based Intervention for Pregnant Women with a Baby in Breech Presentation
Brief Title: Mindfulness-based Intervention Prior to External Cephalic Version
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Tilburg University (Other)
Responsible Party: Principal Investigator, Simone Kuppens, Principal Investigator, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W24.245
Record Dates: First submitted 2024-12-17; First posted 2025-01-10 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Breech Presentation in Pregnancy; External Cephalic Version
Keywords: Breech presentation; Pregnancy; External cephalic version; Mindfulness intervention
MeSH Terms: conditions — Breech Presentation

STUDY DESIGN:
Intervention Model Description: Randomization stratified for parity.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Short mindfulness-based intervention (5 minutes) prior to the external cephalic version
  Interventions: Behavioral: Short mindfulness-based intervention
- Control group (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Short mindfulness-based intervention — The intervention includes a short mindfulness-based intervention with a duration of 5 minutes. It involves a sitting mediation focused on breath adapted from the existing protocols of the Mindfulness-Based Stress Reduction (MBSR) and Mindfulness-Based Cognitive Therapy (MBCT). The intervention is audio-guided and will be delivered via headphones.
  Arms: Intervention group

SUMMARY:
The study is a randomized controlled trial examining the effectiveness of a short mindfulness-based intervention on the success rate of external cephalic version in pregnant women with breech presentation. It is hypothesized that this intervention will increase the ECV success rate and decrease the pain experienced after the ECV.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (18+y).
* With a breech presenting fetus undergoing external cephalic version.
* Dutch/English-speaking or understanding Dutch/English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Post-intervention external cephalic version success rate | 1 hour after enrollment (i.e., in hospital, after intervention and external cephalic version)
  The success rate of the external cephalic versions (successful/not successful) will be compared between the intervention and control group.

SECONDARY OUTCOMES:
Post-intervention pain perception | 1 hour after enrollment (i.e., in hospital, after intervention and external cephalic version)
  The pain experienced during the external cephalic version will be assessed with a visual analogue scale (VAS). The mean/median VAS scores will be compared between the intervention and control group. The scores range between 0 and 10, with a higher score indicating more experienced pain.
Post-intervention comfort | 1 hour after enrollment (i.e., in hospital, after intervention and external cephalic version)
  Comfort during the external cephalic version will be assessed with a visual analogue scale (VAS). The mean/median VAS scores will be compared between the intervention and control group. The scores range between 0 and 10, with a higher score indicating more comfort.

OTHER OUTCOMES:
Baseline mindfulness skills | At baseline (i.e., in hospital, prior to intervention and external cephalic version)
  Baseline mindfulness skills are assessed with the 15-item Three Facet Mindfulness Questionnaire Short Form (TFMQ-SF), consisting of the facets acting with awareness, non-judging and non-reacting. The total score ranges from 0 to 60, with higher scores indicating better mindfulness skills. The validity of the measure is established and indices of internal reliability were found to be adequate.
Baseline depressive symptoms | At baseline (i.e., in hospital, prior to intervention and external cephalic version)
  Assessed with the 10-item Edinburgh Postnatal Depression Scale (EPDS). The EPDS is the most widely used self-rating scale to assess depressive symptoms in the perinatal period. The EPDS total score ranges from 0 to 30, with higher scores indicating more depressive symptoms. The questionnaire has been validated in Dutch postpartum women.
Baseline fear of external cephalic version | At baseline (i.e., in hospital, prior to intervention and external cephalic version)
  Assessed with a visual analogue skill (VAS), by which participants indicate how anxious they feel about the upcoming external cephalic version. The scores range from 0 to 10, with higher scores indicating more anxiety about the upcoming external cephalic version.
Post-intervention general questions | 1 hour after enrollment (i.e., in hospital, after intervention and external cephalic version)
  Three general questions about the information that women received during the external cephalic version, and the familiarity with mindfulness/yoga.
Post-intervention evaluation of the intervention | 1 hour after enrollment (i.e., in hospital, after intervention and external cephalic version)
  Four questions about how women perceived the intervention (intervention group only)

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands